CLINICAL TRIAL: NCT02141750
Title: THIRD NATIONAL REGISTRY OF ACUTE CORONARY SYNDROMES
Acronym: RENASICA_III
Status: Completed | Type: Observational
Sponsor: Third National Registry of Acute Coronary Syndromes (Other)
Responsible Party: Sponsor
Other Study IDs: RENASICA III
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Registry pretends to identify stratification, diagnosis and treatment approaches in patients with Acute Coronary Syndrome (ACS) in community hospitals with tertiary hospitals to optimize resources and identify strategies to improve health care quality through the creation of clinical guidelines that serve for unify management and treatment methods with adherence to international guidelines which include suggestions for treatment and medication.

ELIGIBILITY:
Inclusion Criteria:

all patients with suspected ACS and will analyze risk factors, chest pain and electrocardiographic characteristics.

Exclusion Criteria:

Patients with secondary ischemia (anaemia, pulmonary thromboembolism, myocarditis) and type II infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will include patients older than 18 years with ACS final diagnosis and objective evidence of atherosclerotic coronary disease. Patients will be identified in the emergency department, coronary care units, intensive care units, hospital and hemodynamic laboratories
Sampling Method: Probability Sample
Enrollment: 8296 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with complications after presenting ACS | up to one year
  The main objective will be to know the evolution of ACS in third and second level hospitals with a monitoring at a minimum of one year for each patient.